CLINICAL TRIAL: NCT07093931
Title: A Phase Ⅲ Study to Evaluate Efficacy and Safety of Lobaplatin and Carboplatin as Neoadjuvant Therapy in Participants With HER-2 Positive Breast Cancer.
Brief Title: Efficacy and Safety of Lobaplatin and Carboplatin as Neoadjuvant Therapy in HER-2 Positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science (Unknown)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-III-HER2+-001
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: HER-2 positive breast cancer; Pathological Complete Response; Neoadjuvant Therapt; lobaplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — lobaplatin; Carboplatin; Docetaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel or albumin paclitaxel+carboplatin+Trastuzumab+pertuzumab (Other): Docetaxel ( 75 mg / m2 i.v. d1, q3w ) or albumin paclitaxel ( 260 mg / m2 i.v. d1, q3w ) combined with carboplatin ( AUC 5-6 i.v. q3w ) for 6 cycles. Trastuzumab combined with pertuzumab : 6 cycles of treatment, according to the instructions recommended dosage.
  Interventions: Drug: carboplatin; Drug: Docetaxel or albumin paclitaxel; Drug: Trastuzumab; Drug: pertuzumab
- Docetaxel or albumin paclitaxel+lobaplatin +Trastuzumab+pertuzumab (Experimental): Docetaxel ( 75mg / m2 i.v. d1, q3w ) or albumin paclitaxel ( 260mg / m2 i.v. d1, q3w ) combined with lobaplatin ( 30mg / m2 i.v. q3w ) for 6 cycles. Trastuzumab combined with pertuzumab : 6 cycles of treatment, according to the instructions recommended dosage.
  Interventions: Drug: lobaplatin; Drug: Docetaxel or albumin paclitaxel; Drug: Trastuzumab; Drug: pertuzumab

INTERVENTIONS:
Drug: lobaplatin — 30mg / m2 i.v. q3w
  Arms: Docetaxel or albumin paclitaxel+lobaplatin +Trastuzumab+pertuzumab
Drug: carboplatin — AUC 5-6 i.v. q3w
  Arms: Docetaxel or albumin paclitaxel+carboplatin+Trastuzumab+pertuzumab
Drug: Docetaxel or albumin paclitaxel — Docetaxel ( 75 mg / m2 i.v. d1, q3w ) or albumin paclitaxel ( 260 mg / m2 i.v. d1, q3w )
Drug: Trastuzumab — 6 cycles of treatment, according to the instructions recommended dosage.
Drug: pertuzumab — 6 cycles of treatment, according to the instructions recommended dosage.

SUMMARY:
The aim of this study was to evaluate the efficacy, safety and tolerability of lobaplatin versus carboplatin as neoadjuvant therapy for stage II / III HER-2 positive breast cancer.

Arms and Interventions Control group : Docetaxeor albumin paclitaxel combined with carboplatin for 6 cycles. Trastuzumab combined with pertuzumab : 6 cycles of treatment, according to the instructions recommended dosage.

Experimental group : Docetaxel or albumin paclitaxel combined with lobaplatin for 6 cycles. Trastuzumab combined with pertuzumab : 6 cycles of treatment, according to the instructions recommended dosage.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer
* 18-70 Years, female;
* life expectancy is not less than 3 months
* Histologically confirmed HER2 positive ( human epidermal growth factor receptor 2 [ HER2 ] positive, estrogen receptor [ ER ] and progesterone receptor [ PR ] negative or positive );
* Stage at presentation: T1c N1-2 or T2-4 N0-2;
* at least one measurable lesion according to RECIST 1.1;

Adequate function of major organs meets the following requirements:

* Neutrophils ≥ 1.5×10^9/L
* Platelets ≥ 100×10^9/L
* Hemoglobin ≥ 90g/L
* lymphocyte≥0.5×10^9/L
* Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
* ALT and AST ≤ 3 × ULN
* ALP≤ 2.5 × ULN
* BUN and Cr ≤ 1.5 × ULN
* TSH≤ ULN
* Left ventricular ejection fraction (LVEF) ≥ 50%
* QTcF ≤ 470 ms
* Provides tumor tissue specimen to assess tumor programmed death-ligand 1 (PD-L1); .For women of childbearing potential: agreement to use contraceptive methods. Women who are not postmenopausal or have undergone a sterilization procedure must have a negative serum pregnancy test result within 72 hours prior to initiation of study drug.

Exclusion Criteria:

* Stage Ⅳ (metastatic) breast cancer or bilateral breast cancer
* Inflammatory breast cancer
* patients who received chemotherapy, endocrine therapy, immunotherapy, biotherapy or TACE within 4 weeks before admission
* Has participated in an interventional clinical study with an investigational compound within 4 weeks prior to initiation of study treatment
* Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies .Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Major surgical procedure within 4 weeks prior to initiation of study treatment
* Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus
* Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases
* Administration of a live attenuated vaccine within 28 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study .Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B, Hepatitis C or Autoimmune hepatitis
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment
* Has evidence of active tuberculosis within 1year prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Pre-existing motor or sensory neuropathy of a severity≥grade 2
* Has significant cardiovascular disease
* Treatment with systemic immunostimulatory agents within 4 weeks prior to initiation of study treatment
* Treatment with systemic immunosuppressive medications within 2 weeks prior to initiation of study treatment
* Has a known hypersensitivity to the components of the study treatment or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial .History of neurological or psychiatric disorders, including epilepsy or dementia.
* any other situation evaluated by researchers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive tumor on hematoxylin and eosin evaluation of breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.
Adverse events (AEs) | Up to approximately 35 weeks
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

SECONDARY OUTCOMES:
Event-Free Survival (EFS) in all participants | Up to approximately 5 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Objective Overall Response Rate (ORR) | Up to approximately 25-30 weeks
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until definitive surgery or disease progression.
Disease-free survival ( DFS ) | Up to approximately 5 years
  DFS is defined as the time interval from the first day of disease-free ( i.e., the date of surgery ) to the first recording of related events, including postoperative disease recurrence and metastasis and death from any cause.
Distant Disease-Free Survival(DDFS) | Up to approximately 5 years
  DDFS is defined as the time interval from the beginning of treatment ( such as surgery, radiotherapy or drug intervention ) to the first occurrence of distant metastasis or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Cancer Center Shandong Cancer Hospital and Institute Shandong First Medical University and Shandong Academy of Medical Sciences, Shandong, Jinan, China

IPD SHARING:
Plan to Share IPD: Yes